CLINICAL TRIAL: NCT05800535
Title: Prevalence of Sarcopenia and Chemobrain in Post-cancer Patients
Brief Title: JUMP Prevalence of Sarcopenia and Chemobrain in Post-cancer Patients
Acronym: JUMP
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 813; 69HCL23_0177 (Other: HCL)
Record Dates: First submitted 2023-03-24; First posted 2023-04-05 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Cancer; Sarcopenia
Keywords: Post cancer; Chemobrain; Sarcopenia; Medical evaluation
MeSH Terms: conditions — Neoplasms; Sarcopenia; Chemotherapy-Related Cognitive Impairment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- JUMP Cohort: This study concerns adults with cancer treated with chemotherapy, radiotherapy, hormonal therapy or immunotherapy, in remission or cured. Patients took part in the dedicated post-cancer assessment day.
  Interventions: Drug: Study of the adverse effects of long-term oncological treatments; Behavioral: Study of the long-term side effects of oncological treatments on the anxiety-depressive and cognitive state of patients

INTERVENTIONS:
Drug: Study of the adverse effects of long-term oncological treatments — Cognitive and muscular evaluation of patients who have received oncological treatments, away from the latest treatments to assess their impacts
Behavioral: Study of the long-term side effects of oncological treatments on the anxiety-depressive and cognitive state of patients — Cognitive and anxiety-depressive evaluation of patients who have received oncological treatments, away from the latest treatments to assess their impacts

SUMMARY:
Therapeutic advances in oncology have transformed the prognosis of cancer patients, placing a significant number of them either in a context of recovery or in prolonged remission close to a chronic disease. Thus, the reconquest of a life after cancer becomes possible but raises many challenges for the patient, his entourage, the medical profession and our society. One of the major challenges is the detection and management of treatment side effects for all patients. In addition to the standard organic assessment (glycaemia, creatinine, liver test, blood count), we are mainly interested in muscle deconditioning and cognitive impairment, which are particularly disturbed in these populations. After the evaluation day, patients are referred to the most appropriate structures (Adapted physical activity, sports for health, and rehabilitation at Henry Gabriel Hospital).

JUMP research is part of axis 2 of the 2021-2030 cancer plan: "Limiting sequelae and improving quality of life", through sheets 1 (research) / 6 (access and quality) / 7 (prevention). This leads to the concrete implementation on the territory of adapted care channels in the city: medical structure, physiotherapy, Adapted Physical Activity (APA) structures, associative structures; which makes it possible to develop and strengthen the city-hospital link. Finally, it allows the patient to take ownership and get involved in the project, allowing in the future to make them truly active in they care and to advise and motivate their peers.

This study is non-interventional, it uses research on data that is already collected as part of conventional care, during the JUMP evaluation day.

This study allows the investigators to constitute a cohort of patients to study different parameters related to the disease or to the treatments received.

Our main objective in this study is to describe the muscular and neurocognitive impairment of post-cancer patients evaluated as part of the JUMP program.

ELIGIBILITY:
Inclusion Criteria:

* Age : 18 to 74 years
* localization of the primitive: breast, lung, melanoma, testicle, bladder, kidney, ovary, colon and pancreas, hemopathy
* patient who benefited from the post-cancer assessment day-

Exclusion Criteria:

* Under 18years
* Over 74 years
* Patient who did not received any chemical treatment
* Patient who do not wish to participate

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who have been treated for cancer and who have completed the post-cancer assessment day
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2029-02-10 (Estimated); Study Completion 2029-02-10 (Estimated)

PRIMARY OUTCOMES:
Prevalence of patients with physical and neurocognitive impairment | at least 1 year later after chemical treatments
  Number of patients whose medical assessments show altered physical, cognitive or anxiety/dpression activity compared to the measurement in the general population

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Rhumatologie, Hospices Civils de Lyon, Groupement Hospitalier Lyon Sud, Pierre-Bénite, France